CLINICAL TRIAL: NCT04777864
Title: Developing a Tool to Support Shared Decision Making Post-Concussion Between Adolescents, Parents and Clinicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Emily Kroshus, Research Assistant Professor, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00002334
Record Dates: First submitted 2021-02-23; First posted 2021-03-02 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Concussion, Brain
MeSH Terms: conditions — Brain Concussion | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention)
- Decision Aid (Experimental): Usual care, plus introduction of a decision aid
  Interventions: Behavioral: Decision Aid

INTERVENTIONS:
Behavioral: Decision Aid — In addition to usual care, participants (parents and adolescents) receive the newly developed decision aid prior to their clinic visit(s). Clinicians receive a summary to review and use to help facilitate the decision making process.
  Arms: Decision Aid

SUMMARY:
Investigators will conduct a pilot efficacy test of a decision aid about contact sport participation post-concussion.

DETAILED DESCRIPTION:
The clinical trial portion of this study will enroll 40 adolescents and their parent/caregiver who are seen in the Sports Medicine clinic with a diagnosis of concussion. 20 will receive usual care, and 20 will receive a decision aid to facilitate the decision making process about sport participation post-concussion. Adolescents and their parent/caregiver will complete separate surveys at a minimum of three timepoints: before their initial clinic visit, after each clinic visit (up until a decision regarding sports participation post-concussion is made), and three months after their first clinic visit. The study team will also conduct surveys with clinicians about their experiences with implementation.

ELIGIBILITY:
Participants in the clinical trial component of this study will be adolescents, parents, and healthcare providers:

Adolescent Inclusion Criteria:

* Age 11-17
* Sustained at least 1 concussion and is scheduled for a concussion injury visit

Parent Inclusion Criteria:

* Age 18 or older
* Parent of a child between the age of 11 and 17 (inclusive) who has sustained at least 1 concussion and is scheduled for a concussion injury visit

Healthcare Provider Inclusion Criteria:

* Age 18 or older
* Seattle Children's affiliated healthcare provider who provides patient care to youth with concussion

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited a sample of adolescents (ages 11-17) and their parent/caregiver who were seen in the Sports Medicine clinic with a diagnosis of concussion. After dyads enrolled, the parent or guardian and adolescent were emailed and/or texted separate surveys to complete before the upcoming appointment.
Pre-assignment Details: All participants were assigned to the control or intervention condition. There were 10 dyads (n=20 participants) enrolled in the intervention that did not complete the intervention prior to their index visit. These dyads were excluded from analyses. 24 dyads (48 participants) were included in the control condition and 21 dyads (42 participants) were included in the intervention condition. The protocol enrollment number represents the number of individual participants enrolled in each condition.
Groups:
- Usual Care: Participants received post-concussion care as usual.
Period: Overall Study
Arm/Group | Usual Care | Decision Aid
Started | 48 (Footnote 1: Started Usual Care: Parents/Guardians=24, Adolescents=24) | 62 (Footnote 2: Decision Aid: Parents/Guardians=31, Adolescents=31)
Index Visit | 45 (Footnote 3: Usual Care T2 Survey Complete: Parents/Guardians=24, Adolescents=21) | 51 (Footnote 4: Decision Aid T2 Survey Complete: Parents/Guardians=26, Adolescents=25)
Completed | 40 (Footnote 5: Usual Care T3 Survey Complete: Parents/Guardians=22, Adolescents=18) | 43 (Footnote 6: Decision Aid T3 Survey Complete: Parents/Guardians=23, Adolescents=20)
Not Completed | 8 | 19
Not completed — Lost to Follow-up | 8 | 19

BASELINE CHARACTERISTICS:
Population: 24 dyads were in the control phase and 46 individual participants (adolescents: n=22; parents: n=24) completed baseline surveys. Of the 31 dyads in the intervention phase, only 21 dyads completed the tool before their index visit and were therefore included in the analyses reported here; the remaining 10 dyads did not complete the tool in time and were excluded. Among the included dyads, 42 individual participants (adolescents: n= 21; parents: n=21) also completed baseline surveys.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Decision Aid | Total
Number analyzed (Participants) | 46 | 42 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data is reported only for individuals who were included in the analyses and responded to this question. Data is reported separately for parents and adolescents.
  years
    Parent: number analyzed (Participants) | 19 | 21 | 40
    Parent | 47.11 (4.61) | 46.05 (3.90) | 46.55 (4.23)
    Adolescent: number analyzed (Participants) | 21 | 21 | 42
    Adolescent | 15.56 (1.40) | 15.59 (1.75) | 15.57 (1.55)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Data is reported only for individuals who were included in the analyses and responded to this question. Data is reported separately for parents and adolescents.
  Participants
    Parent: number analyzed (Participants) | 22 | 21 | 43
    Parent: Female | 14 | 19 | 33
    Parent: Male | 8 | 2 | 10
    Parent: Non-binary | 0 | 0 | 0
    Adolescent: number analyzed (Participants) | 22 | 21 | 43
    Adolescent: Female | 12 | 11 | 23
    Adolescent: Male | 9 | 10 | 19
    Adolescent: Non-binary | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data is reported separately for parents and adolescents.
  Participants
    Parent: number analyzed (Participants) | 24 | 21 | 45
    Parent: Hispanic or Latino | 1 | 1 | 2
    Parent: Not Hispanic or Latino | 21 | 20 | 41
    Parent: Unknown or Not Reported | 2 | 0 | 2
    Adolescent: number analyzed (Participants) | 22 | 21 | 43
    Adolescent: Hispanic or Latino | 1 | 3 | 4
    Adolescent: Not Hispanic or Latino | 21 | 18 | 39
    Adolescent: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data is reported separately for parents and adolescents.
  Participants
    Parent: number analyzed (Participants) | 24 | 21 | 45
    Parent: American Indian or Alaska Native | 0 | 0 | 0
    Parent: Asian | 2 | 1 | 3
    Parent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parent: Black or African American | 1 | 0 | 1
    Parent: White | 19 | 19 | 38
    Parent: More than one race | 0 | 0 | 0
    Parent: Unknown or Not Reported | 2 | 1 | 3
    Adolescent: number analyzed (Participants) | 22 | 21 | 43
    Adolescent: American Indian or Alaska Native | 0 | 0 | 0
    Adolescent: Asian | 2 | 0 | 2
    Adolescent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Adolescent: Black or African American | 2 | 0 | 2
    Adolescent: White | 18 | 20 | 38
    Adolescent: More than one race | 0 | 0 | 0
    Adolescent: Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Decisional Regret
Description: We used the 5-item Decisional Regret Scale to measure personal perceptions of regret when considering the decision previously made about sports participation post-concussion. Responses are on a 5-point Likert scale, from (1) strongly agree to (5) strongly disagree. Two positively worded items were reverse scored. Responses were averaged to create a decisional regret score with a possible range of 1 to 5, with higher scores indicating greater regret.
Time Frame: 3 months after initial clinic visit
Population: The number analyzed in one or more rows differs from the overall number analyzed because only participants who completed the scale at 3-month follow-up survey were included in the analyses. Outcomes are also reported separately by subgroup (parent, child).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Usual Care | Decision Aid
Number analyzed (Participants) | 41 | 36
Score on a scale
  Parents: number analyzed (Participants) | 22 | 18
  Parents | 1.68 (0.64) | 2.00 (0.83)
  Adolescents: number analyzed (Participants) | 19 | 18
  Adolescents | 1.80 (1.09) | 1.77 (0.69)
Statistical Analysis 1: Comparison: Usual Care vs Decision Aid; Parent group only; Test type: Superiority; p = 0.18, t-test, 2 sided
Statistical Analysis 2: Comparison: Usual Care vs Decision Aid; Adolescent group only; Test type: Superiority; p = 0.91, t-test, 2 sided

2. Primary Outcome: Change in Quality of Choice Made
Description: We used the 10-item Decisional Conflict Scale-Low Literacy version to measure parent and adolescent perceptions of certainty in making the decision to return to sports after concussion recovery. Respondents answered 10 items using a 3-point scale scored as 0 = "yes," 2 = "unsure," and 4 = "no." Item scores were summed, divided by 10, and then multiplied by 25 to produce a total decisional conflict score ranging from 0 to 100, with higher scores indicating greater decisional conflict and lower decision certainty.
Time Frame: Baseline: Within 1 week prior to the index clinic visit (i.e., the participant's first visit after they enrolled in the study), Post-Index Visit: Within 24 hours after the index visit (typically occurs 1-2 weeks after enrollment),
Population: The number analyzed in one or more rows differs from the overall number because results are reported separately by group (Parent, Child) and timepoint (Baseline, Post-Index Visit). The number reported for each timepoint includes only those participants who responded at that timepoint and, for the Post-Index Visit timepoint, also reported that they made a decision.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Usual Care | Decision Aid
Number analyzed (Participants) | 44 | 42
Score on a scale
  Parent: Baseline: number analyzed (Participants) | 21 | 21
  Parent: Baseline | 43.81 (18.43) | 42.62 (21.83)
  Adolescent: Baseline: number analyzed (Participants) | 22 | 21
  Adolescent: Baseline | 20.91 (21.02) | 20.95 (26.06)
  Parent: Post-Index Visit: number analyzed (Participants) | 23 | 21
  Parent: Post-Index Visit | 15.00 (19.31) | 13.81 (16.87)
  Adolescent: Post-Index Visit: number analyzed (Participants) | 21 | 20
  Adolescent: Post-Index Visit | 7.62 (18.07) | 7.75 (13.81)
Statistical Analysis 1: Comparison: Usual Care vs Decision Aid; Parent: Post-Index Visit; Test type: Superiority; p = 0.975, Regression, Linear
Statistical Analysis 2: Comparison: Usual Care vs Decision Aid; Adolescent: Post-Index Visit; Test type: Superiority; p = 0.854, Regression, Linear

3. Primary Outcome: Decision Self-Efficacy
Description: We used a 12-item Decision Self-Efficacy Scale to measure parent and adolescent confidence in making health-related decisions. Participants responded using a 5-point scale scored from 0 = "not at all confident" to 4 = "very confident." Item scores were summed, divided by 12, and then multiplied by 25 to produce a total decision self-efficacy score ranging from 0 to 100, with higher scores indicating greater confidence in decision-making. The scale included an additional item: "Let my child/my parent(s) know what I think is best for them/me."
Time Frame: Baseline: Within 1 week prior to the index clinic visit (i.e., first visit after enrolled in the study)
Population: The number analyzed in one or more rows differs from the overall number because results are reported separately by group (Parent, Adolescent).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Decision Aid
Number analyzed (Participants) | 40 | 40
score on a scale
  Parent: number analyzed (Participants) | 20 | 20
  Parent | 80.41 (15.09) | 77.29 (17.62)
  Adolescent: number analyzed (Participants) | 20 | 20
  Adolescent | 77.91 (14.01) | 79.90 (17.17)

4. Primary Outcome: Patient-Parent-Provider Engagement
Description: We used the 19-item Decision Making Involvement Scale to assess engagement and perceived support in the decision making process, divided into two subscales: Within Family Engagement and Family-Provider Engagement. Participants rated their agreement with items on a 4-point Likert scale from 1 (strongly disagree) to 4 (strongly agree). Subscale scores are calculated by averaging the item responses within each subscale. Each subscale score ranges from 1 to 4, with higher scores indicating more engagement or involvement.
Time Frame: Post-Index Visit: Within 24 hours after the index visit (typically occurs 1-2 weeks after enrollment),
Population: Analyses only include participants who reported that they made a decision after their first visit. Outcomes are reported separately by subgroup (parent, child) and subscale (within family engagement and family-clinician engagement).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Decision Aid
Number analyzed (Participants) | 22 | 20
score on a scale
  Parent: Within family engagement: number analyzed (Participants) | 10 | 11
  Parent: Within family engagement | 2.83 (0.60) | 2.76 (0.55)
  Adolescent: Within family engagement: number analyzed (Participants) | 11 | 9
  Adolescent: Within family engagement | 2.68 (0.84) | 3.07 (0.49)
  Parent: Family-clinician engagement: number analyzed (Participants) | 11 | 11
  Parent: Family-clinician engagement | 2.94 (0.43) | 2.87 (0.55)
  Adolescent: Family-clinician engagement: number analyzed (Participants) | 11 | 10
  Adolescent: Family-clinician engagement | 3.20 (0.36) | 3.25 (0.39)

5. Secondary Outcome: Change in Adolescent Physical Activity
Description: We used the International Physical Activity Questionnaire (IPAQ-SF) to assess adolescent physical activity post-concussion. Participants reported the number of days and minutes spent on vigorous, moderate, and walking activities. These values were converted to MET-minutes per week (MMW) using standard MET values (vigorous = 8, moderate = 4, walking = 3.3). The total physical activity score was calculated by summing the MMW for all activities.
Time Frame: Baseline: Within 1 week prior to the index clinic visit (i.e., first visit after enrolled in the study), Post-Index Visit: Within 24 hours after the index visit (typically occurs 1-2 weeks after enrollment), 3 months after initial clinic visit
Population: The number analyzed in one or more rows differs from the overall number because these analyses include only adolescent participants.
Measure: Mean (Standard Deviation); unit: total mmw
Arm/Group | Usual Care | Decision Aid
Number analyzed (Participants) | 21 | 21
total mmw
  Post-Index Visit | 466 (581.02) | 1220.79 (1440.68)
  3 Month Follow-up: number analyzed (Participants) | 18 | 18
  3 Month Follow-up | 2141.39 (1111.35) | 1775.11 (1378.90)
Statistical Analysis 1: Comparison: Usual Care vs Decision Aid; Post-Index Visit; Test type: Superiority; p = 0.03, t-test, 2 sided
Statistical Analysis 2: Comparison: Usual Care vs Decision Aid; 3 months after initial clinic visit; Test type: Superiority; p = 0.21, t-test, 2 sided

6. Secondary Outcome: Change in Adolescent Psychosocial Functioning
Description: We used the Pediatric Quality of Life Inventory, Psychosocial subscale (PEDS-QL) to measure adolescent emotional functioning. Participants rated items on a 5-point Likert scale, with higher scores reflecting better emotional functioning. To ensure ease of interpretation, items were reverse scored and then transformed to a 0-100 scale, where higher scores indicate better emotional health.
Time Frame: as for outcome 5
Population: The number analyzed in one or more rows differs from the overall number because results are reported separately by timepoint (Baseline, Post-Index Visit, 3 Month Follow-up). The number reported for each timepoint includes only those participants who responded at that timepoint .
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Usual Care | Decision Aid
Number analyzed (Participants) | 22 | 21
Score on a scale
  Baseline | 81.14 (16.10) | 79.52 (18.43)
  Post-Index Visit: number analyzed (Participants) | 21 | 21
  Post-Index Visit | 84.05 (14.97) | 83.81 (15.56)
  3-Month Follow-up: number analyzed (Participants) | 21 | 21
  3-Month Follow-up | 84.05 (14.96) | 83.81 (15.56)
Statistical Analysis 1: Comparison: Usual Care vs Decision Aid; Baseline; Test type: Superiority; p = 0.76, t-test, 2 sided
Statistical Analysis 2: Comparison: Usual Care vs Decision Aid; Post-Index Visit; Test type: Superiority; p = 0.96, t-test, 2 sided
Statistical Analysis 3: Comparison: Usual Care vs Decision Aid; 3 months after initial clinic visit; Test type: Superiority; p = 0.96, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- Usual Care - Parents; Usual Care - Adolescents: Participants received post-concussion care as usual.
- Decision Aid - Parents; Decision Aid - Adolescents: Usual care, plus introduction of a decision aid
  Decision Aid: In addition to usual care, participants (parents and adolescents) receive the newly developed decision aid prior to their clinic visit(s). Clinicians receive a summary to review and use to help facilitate the decision making process.
Arm/Group | Usual Care - Parents | Decision Aid - Parents | Usual Care - Adolescents | Decision Aid - Adolescents
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21 | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21 | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21 | 0/24 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT04777864/Prot_SAP_000.pdf
  • Informed Consent Form: Control Group (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT04777864/ICF_001.pdf
  • Informed Consent Form: Intervention Group (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/64/NCT04777864/ICF_002.pdf